CLINICAL TRIAL: NCT01881776
Title: Continuous Interscalene Block in Patients Having Outpatient Rotator Cuff Repair Surgery: a Prospective Randomized Trial
Brief Title: Continuous Interscalene Block Results in Superior Recovery Throughout the First Postoperative Week
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10142
Record Dates: First submitted 2013-02-26; First posted 2013-06-20 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2013-07

CONDITIONS: Postoperative Pain; Adverse Effects
Keywords: Single injection interscalene brachial plexus block; Continuous interscalene brachial plexus block; General anesthesia; Postoperative pain; Recovery profile
MeSH Terms: conditions — Pain, Postoperative | interventions — Catheters

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Single ISB (SISB) group (Active Comparator): Patients in this group received single injection (SISB) interscalene brachial plexus block
  Interventions: Procedure: ISB
- Continuous ISB (CISB) group (Active Comparator): Patients in this group received continuous (CISB) interscalene brachial plexus block
  Interventions: Procedure: ISB
- General anesthesia (GA) group (No Intervention): Patients in this group received general anesthesia (GA)

INTERVENTIONS:
Procedure: ISB — In SISB group; a 5 cm block needle (Stimuplex®A, B Braun Medical, Bethlehem, PA) was inserted in-plane in order to place the needle tip between the upper and middle trunks of the brachial plexus (C5-C6). 20 mL 0.5% ropivacaine was injected through the needle.
  For CISB, a 5cm stimulating needle (Contiplex® Tuohy, B. Braun Medical, Bethlehem, PA) was inserted in-plane in order to place the needle tip between the upper and middle trunks of the brachial plexus (C5-C6). A nonstimulating catheter was inserted approximately 3 cm beyond the tip of the needle. 20 mL 0.5% ropivacaine was injected through the catheter.
  Other Names: SISB needle (Stimuplex®A, B Braun); CISB needle and catheter (Contiplex® Tuohy, B. Braun)
  Arms: Continuous ISB (CISB) group; Single ISB (SISB) group

SUMMARY:
The investigators undertook this prospective, randomized trial to compare the recovery profile throughout the first postoperative week in patients receiving continuous (CISB) interscalene brachial plexus block, single injection (SISB), or general anesthesia (GA) for arthroscopic rotator cuff repair surgery. Specifically, the effects of the three anesthetic techniques when used intraoperatively as a sole anesthesia modality were studied on postoperative pain, time-to-first pain, analgesic consumption, fast-tracked PACU bypass rate, length of PACU stay, time-to-discharge home, sleep duration, and related adverse effects. The investigators hypothesized that CISB results in a superior postoperative recovery profile as compared to SISB or GA alone.

DETAILED DESCRIPTION:
Background The advantages of single injection (SISB) and continuous interscalene brachial plexus block (CISB) over general anesthesia (GA) only have been previously reported. However, few studies extended their observations beyond 48 postoperative hours, and no study has compared the effects of SISB and CISB as sole anesthesia modalities with GA only. We undertook this randomized trial to compare the recovery profile of patients receiving SISB, CISB or GA for arthroscopic rotator cuff repair surgery through the first postoperative week. Our primary hypothesis was that highest NRS pain rating (worst pain score) at the end of the study week is lower for patients in the CISB group than for patients in the SISB or GA groups.

Methods After Institutional Review Board approval and informed consents were obtained, 71 patients of American Society of Anesthesiologists (ASA) physical status I-III, ≥18 years of age, and BMI≤35 kg/m2, scheduled for elective outpatient arthroscopic rotator cuff repair, were enrolled. CISB patients received 20 mL of 0.5% ropivacaine as bolus through the catheter whereas SISB patients received the same volume of injection through a needle. CISB patients received an infusion of 0.2% ropivacaine at 5mL/h with a patient controlled bolus of 5 mL hourly. GA only patients received a standardized general anesthetic. All patients were prescribed acetaminophen (500mg) with hydrocodone (7.5mg) every 4h as needed. CISB was discontinued 48 h after surgery. Postoperative highest pain scores (NRS) through the first postoperative week, time-to-first pain, analgesic consumption, fast-tracked postoperative care unit (PACU) bypass rate, length of PACU stay, time-to-discharge home, sleep duration, and related adverse effects were recorded in the PACU and at home on postoperative days 1, 2, 3, and 7.

ELIGIBILITY:
Inclusion Criteria:

American Society of Anesthesiologists (ASA) physical status I-III patients

≥ 18 years of age BMI ≤ 35 kg/m2 Scheduled for elective arthroscopic shoulder surgery

Exclusion Criteria:

Patients who were undertaken open shoulder procedures Patients with difficulty understanding the instructions for using the anesthetic infusion pump and/or pain scales Patients with contraindications to regional anesthesia (e.g., allergy to a local anesthetic (LA), local infection, coagulopathy) Patients with significant neurologic disorders of the upper extremity, psychiatric or cognitive disorders, history of substance abuse or chronic opioid use

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Admir Hadzic, MD,PhD,Prof, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- St Luke's Roosevelt Hospital Center, New York, New York, United States

REFERENCES:
- [Derived] Salviz EA, Xu D, Frulla A, Kwofie K, Shastri U, Chen J, Shariat AN, Littwin S, Lin E, Choi J, Hobeika P, Hadzic A. Continuous interscalene block in patients having outpatient rotator cuff repair surgery: a prospective randomized trial. Anesth Analg. 2013 Dec;117(6):1485-92. doi: 10.1213/01.ane.0000436607.40643.0a. PMID 24257398
- See also: SINGLE INJECTION ISB — http://www.nysora.com/peripheral_nerve_blocks/ultrasound-guided_techniques/3328-us-guided-interscalene-brachial-plexus-block.html
- See also: CONTINUOUS ISB — http://www.nysora.com/peripheral_nerve_blocks/ultrasound-guided_techniques/3329-ultrasound-guided-continuous-interscalene-block.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: St Luke's-Roosevelt Hospital Center between August 2011 and June 2012
Pre-assignment Details: One patient enrolled preferred to get SISB instead of GA and was therefore not randomized to treatment.
Groups:
- Single ISB (SISB) Group: Patients in this group received single injection (SISB) interscalene brachial plexus block
  ISB : In SISB group; a 5 cm block needle (Stimuplex®A, B Braun Medical, Bethlehem, PA) was inserted in-plane in order to place the needle tip between the upper and middle trunks of the brachial plexus (C5-C6). 20 mL 0.5% ropivacaine was injected through the needle.
  For CISB, a 5cm stimulating needle (Contiplex® Tuohy, B. Braun Medical, Bethlehem, PA) was inserted in-plane in order to place the needle tip between the upper and middle trunks of the brachial plexus (C5-C6). A nonstimulating catheter was inserted approximately 3 cm beyond the tip of the needle. 20 mL 0.5% ropivacaine was injected through the catheter.
- Continuous ISB (CISB) Group: Patients in this group received continuous (CISB) interscalene brachial plexus block
  ISB : In SISB group; a 5 cm block needle (Stimuplex®A, B Braun Medical, Bethlehem, PA) was inserted in-plane in order to place the needle tip between the upper and middle trunks of the brachial plexus (C5-C6). 20 mL 0.5% ropivacaine was injected through the needle.
  For CISB, a 5cm stimulating needle (Contiplex® Tuohy, B. Braun Medical, Bethlehem, PA) was inserted in-plane in order to place the needle tip between the upper and middle trunks of the brachial plexus (C5-C6). A nonstimulating catheter was inserted approximately 3 cm beyond the tip of the needle. 20 mL 0.5% ropivacaine was injected through the catheter.
Period: Overall Study
Arm/Group | Single ISB (SISB) Group | Continuous ISB (CISB) Group | General Anesthesia (GA) Group
Started | 24 | 24 | 22
Completed | 23 | 20 | 20
Not Completed | 1 | 4 | 2
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Protocol Violation | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single ISB (SISB) Group | Continuous ISB (CISB) Group | General Anesthesia (GA) Group | Total
Number analyzed (Participants) | 24 | 24 | 22 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 19 | 58
  >=65 years | 5 | 4 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (9) | 56 (10) | 52 (12) | 55 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 14 | 44
  Male | 11 | 7 | 8 | 26
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 22 | 70

OUTCOME MEASURES:

1. Primary Outcome: Patients With Pain: Numerical Rating Scale (NRS-11(0-10): 0:no Pain and 10:Severe/Worst Pain) ≥ 4
Description: The effects of the three anesthetic techniques (continuous interscalene brachial plexus block (CISB), single interscalene brachial plexus block (SISB), or general anesthesia (GA)) when used intraoperatively as a sole anesthesia modality were studied on postoperative pain (highest NRS pain rating)
Time Frame: throughout the first postoperative week on days 1, 2, 3, and 7
Measure: Number; unit: participants
Arm/Group | Single ISB (SISB) Group | Continuous ISB (CISB) Group | General Anesthesia (GA) Group
Number analyzed (Participants) | 23 | 20 | 20
participants | 19 [18 to 25] | 5 [18 to 25] | 11 [18 to 25]

2. Secondary Outcome: Time-to-first Pain
Description: The effects of the three anesthetic techniques (SISB, CISB, and GA) when used intraoperatively as a sole anesthesia modality were studied on postoperative pain (time-to-first pain).
Time Frame: throughout the first postoperative week
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Single ISB (SISB) Group | Continuous ISB (CISB) Group | General Anesthesia (GA) Group
Number analyzed (Participants) | 23 | 20 | 20
hours | 11 (5) | 26 (24) | 2 (3)

3. Secondary Outcome: The Number of Patients Consume ≥1 Dose of Analgesics
Description: The effects of the three anesthetic techniques (SISB, CISB, and GA) when used intraoperatively as a sole anesthesia modality were studied on postoperative pain (analgesic consumption).
Time Frame: throughout the first postoperative week
Measure: Number; unit: participants
Arm/Group | Single ISB (SISB) Group | Continuous ISB (CISB) Group | General Anesthesia (GA) Group
Number analyzed (Participants) | 23 | 20 | 20
participants | 16 | 12 | 13

4. Other Pre Specified Outcome: Fast-tracked Postoperative Care Unit (PACU) Bypass Patient Number
Description: To compare the recovery profile of patients receiving CISB, SISB, or GA for arthroscopic rotator cuff repair surgery throughout the first postoperative week by using fast-tracked PACU bypass rate
Time Frame: throughout the first postoperative week (how many patients left PACU immediately just after the operation)
Measure: Number; unit: participants
Arm/Group | Single ISB (SISB) Group | Continuous ISB (CISB) Group | General Anesthesia (GA) Group
Number analyzed (Participants) | 23 | 20 | 20
participants | 20 | 19 | 0

5. Other Pre Specified Outcome: Length of PACU Stay
Description: To compare the recovery profile of patients receiving CISB, SISB, or GA for arthroscopic rotator cuff repair surgery throughout the first postoperative week by using length of PACU stay.
Time Frame: throughout the first postoperative week (how long patients stayed in PACU just after the operation)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Single ISB (SISB) Group | Continuous ISB (CISB) Group | General Anesthesia (GA) Group
Number analyzed (Participants) | 23 | 20 | 20
minutes | 30 (42) | 20 (31) | 165 (118)

6. Other Pre Specified Outcome: Time to Discharge Home
Description: To compare the recovery profile of patients receiving CISB, SISB, or GA for arthroscopic rotator cuff repair surgery throughout the first postoperative week by using time-to-discharge home.
Time Frame: throughout the first postoperative week (how long patients stayed in the hospital (includes PACU and hospital time)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Single ISB (SISB) Group | Continuous ISB (CISB) Group | General Anesthesia (GA) Group
Number analyzed (Participants) | 23 | 20 | 20
minutes | 115 (109) | 94 (55) | 302 (249)

7. Other Pre Specified Outcome: Total Hours of Sleep
Description: To compare the recovery profile of patients receiving CISB, SISB, or GA for arthroscopic rotator cuff repair surgery throughout the first postoperative week by using sleep duration.
Time Frame: first postoperative week (on day 7)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Single ISB (SISB) Group | Continuous ISB (CISB) Group | General Anesthesia (GA) Group
Number analyzed (Participants) | 23 | 20 | 20
hours | 5 (2) | 7 (1) | 6 (2)

ADVERSE EVENTS:
Time Frame: Throughout the first postoperative week
Description: Postoperative Dizziness, Nausea and Vomiting (PONV): All these symptoms were asked altogether to the patients and assessed only as positive or negative
Arm/Group | Single ISB (SISB) Group | Continuous ISB (CISB) Group | General Anesthesia (GA) Group
Serious Adverse Events (participants affected / at risk) | 5/23 | 0/20 | 2/20
Other Adverse Events (participants affected / at risk) | 0/23 | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single ISB (SISB) Group (N=23) | Continuous ISB (CISB) Group (N=20) | General Anesthesia (GA) Group (N=20)
PONV (Gastrointestinal disorders) | 5 (5) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
1. It was difficult to keep three different groups blinded. 2. The resting and mobilization highest/worst NRS pain scores were ignored and only the highest pain scores of the postoperative days 1, 2, 3, and 7 were recorded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No